CLINICAL TRIAL: NCT01416155
Title: A Long-Term, Open-Label, Multicenter, Extension Study to Evaluate Safety and Efficacy of BG00002 in Japanese Subjects With Relapsing-Remitting Multiple Sclerosis
Brief Title: Extension Study to Evaluate Safety and Efficacy of Natalizumab in Japanese Participants With Relapsing-Remitting Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101MS204
Record Dates: First submitted 2011-03-24; First posted 2011-08-12 (Estimated); Results first posted 2016-01-14 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2015-12

CONDITIONS: Relapsing-Remitting Multiple Sclerosis; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Natalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- natalizumab (Experimental): 300 mg intravenous (IV) infusions of natalizumab every 4 weeks until product is approved in Japan or development is discontinued in Japan, whichever comes first.
  Interventions: Drug: natalizumab

INTERVENTIONS:
Drug: natalizumab
  Other Names: Tysabri; BG00002

SUMMARY:
The primary objective of the study is to further evaluate the long-term safety and tolerability profiles of BG00002 (natalizumab) in Japanese participants with relapsing-remitting multiple sclerosis (RRMS). The secondary objective of this study is to further evaluate the long-term efficacy profile of BG00002 in Japanese participants with RRMS.

DETAILED DESCRIPTION:
This is a multicenter, long-term, open-label, extension study in participants who have successfully completed Study 101MS203 (NCT01440101).

ELIGIBILITY:
Key Inclusion Criteria:

* Ability to understand the purpose and risks of the study and provide signed and dated informed consent and any authorizations required by local law.
* Subjects who participated in and completed all protocol-related evaluations through Week 24 of Study 101MS203 (NCT01440101).
* Subjects participating in study 101MS204 (NCT01416155) participated either in the open label pharmacokinetics-pharmacodynamics study or placebo-controlled study of natalizumab 300 mg q4wks (parts A and B of study 101MS203, respectively).
* Subjects of childbearing potential must practice effective contraception during the study and be willing and able to continue contraception for 12 weeks after their last dose of study treatment.
* Must be willing to remain free from concomitant immunosuppressive or immunomodulatory treatment (including interferon beta [IFNβ] and long-term systemic corticosteroids) for the duration of the study.

Key Exclusion Criteria Medical History

* Any significant change in medical history since Study 101MS203 (NCT01440101), including laboratory tests, or current clinically important condition that in the opinion of the Investigator would have excluded the subject's participation in the previous study. The Investigator must re-review the subject's medical fitness for participation and consider diseases that would preclude treatment.
* Subjects from Study 101MS203 (NCT01440101) who discontinued study treatment due to an adverse event.
* Subjects who are determined to be persistently positive for anti-BG0002 antibodies based on prior testing.

Treatment History

* Treatment with any of the following medications between last dose of study treatment in Study 101MS203 (NCT01440101) and the start of this study: intravenous immunoglobulin (IVIg), plasmapheresis, cytapheresis, immunosuppressant medications (e.g., mitoxantrone, azathioprine, cyclophosphamide, methotrexate, cyclosporine, FTY720), immunomodulatory medications (including IFNβ and glatiramer acetate [GA]) total lymphoid irradiation, cladribine, T-cell or T-cell receptor vaccination, any murine protein, any other therapeutic monoclonal antibody, or any 4-aminopyridine or related products.

Miscellaneous

* For female subjects, unless postmenopausal for at least 1 year or surgically sterile (does not include tubal ligation), unwillingness to practice effective contraception, as defined by the Investigator, during the study. Women considering becoming pregnant while on study are to be excluded.
* Female subjects who are currently pregnant or breast feeding, including subjects whose pregnancy test is positive at Week 0.
* Unwillingness or inability to comply with the requirements of this protocol, including the presence of any condition (physical, mental, or social) that is likely to affect the subject's ability to comply with the study protocol.
* Subjects with any other condition, clinical finding, or reason that in the opinion of the Investigator and/or the Sponsor makes the subject unsuitable for enrollment into the study.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2010-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (18):
- Japan (18):
  - Research Site, Chiba, Chiba
  - Research Site, Fukuoka, Fukuoka
  - Research Site, Hiroshima, Hiroshima
  - Research Site, Sapporo, Hokkaido
  - Research Site, Tsukuba, Ibaraki
  - Research Site, Morioka, Iwate
  - Research Site, Yokohama, Kanagawa
  - Research Site, Kyoto, Kyoto
  - Research Site, Sendai, Miyagi
  - Research Site, Niigata, Niigata
  - Research Site, Osaka, Osaka
  - Research Site, Suita, Osaka
  - Research Site, Kawagoe, Saitama
  - Research Site, Tokorozawa, Saitama
  - Research Site, Bunkyo-ku, Tokyo
  - Research Site, Kodaira, Tokyo
  - Research Site, Ōta-ku, Tokyo
  - Research Site, Ube, Yamaguchi

REFERENCES:
- [Derived] Saida T, Kira JI, Kishida S, Yamamura T, Ohtsuka N, Ling Y, Torii S, Lucas N, Kuesters G, Steiner D, Tibung JT; Natalizumab Trial Principal Investigators. Safety and Efficacy of Natalizumab in Japanese Patients with Relapsing-Remitting Multiple Sclerosis: Open-Label Extension Study of a Phase 2 Trial. Neurol Ther. 2017 Jun;6(1):39-55. doi: 10.1007/s40120-016-0059-z. Epub 2016 Dec 5. PMID 27921221

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects who participated in and completed all protocol-related evaluations through Week 24 in Study 101MS203 (NCT01440101) were eligible for this study.
Groups:
- Natalizumab: 300 mg intravenous (IV) infusions of natalizumab open label every 4 weeks
Period: Overall Study
Arm/Group | Natalizumab
Started | 97
Completed | 39
Not Completed | 58
Not completed — Adverse Event | 8
Not completed — Positive for anti-BG00002 antibodies | 2
Not completed — Withdrawal by Subject | 33
Not completed — Investigator decision | 8
Not completed — Other | 7

BASELINE CHARACTERISTICS:
Groups:
- Natalizumab: 300 mg IV infusions of natalizumab open label every 4 weeks
Arm/Group | Natalizumab
Number analyzed (Participants) | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.2 (8.67)
Age, Customized [Number; unit: participants]
  18 to 19 years | 1
  20 to 29 years | 16
  30 to 39 years | 44
  40 to 49 years | 28
  50 to 59 years | 7
  >= 60 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66
  Male | 31

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs), Serious AEs (SAEs), and Discontinuations Due to AEs
Description: An AE was any untoward medical occurrence that did not necessarily have a causal relationship with this treatment. An SAE was any untoward medical occurrence that at any dose: resulted in death; in the view of the Investigators, placed the subject at immediate risk of death (a life-threatening event); however, this did not include an event that, had it occurred in a more severe form, might have caused death; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; resulted in a congenital anomaly/birth defect; any other medically important event that, in the opinion of the Investigators, could have jeopardized the subject or may have required intervention to prevent one of the other outcomes listed in the definition above.
Time Frame: Day 1 through First Follow-Up (12 Weeks After Last Infusion) +/- 7 days. Approximately 62 months
Population: Safety population: all participants who received at least 1 dose of study treatment.
Measure: Number; unit: participants
Arm/Group | Natalizumab
Number analyzed (Participants) | 97
participants
  Participants with an event | 92
  Participants with a moderate or severe event | 52
  Participants with a severe event | 10
  Participants with an event related to study drug | 33
  Participants with an SAE | 29
  Participants with an SAE related to study drug | 7
  Participants discontinuing treatment due to event | 10
  Participants withdrawing from study due to event | 10

2. Primary Outcome: Number of Participants With Serum Antibodies to Natalizumab
Description: Negative is defined as negative for antibodies at all post-baseline results. Transient positivity is defined as only 1 positive result. Persistent positivity is defined as 2 positive results separated by at least 6 to 12 weeks.
Time Frame: Day 1 up to approximately 50 months
Population: Immunogenicity population: all participants who had received at least 1 infusion of BG00002, were negative for BG00002 antibodies at baseline and had at least 1 nonmissing post-baseline assessment of antibody status.
Measure: Number; unit: participants
Arm/Group | Natalizumab
Number analyzed (Participants) | 96
participants
  Participants negative | 91
  Participants positive at any time | 5
  Participants transiently positive | 3
  Participants positive at final evaluation only | 2
  Participants persistently positive | 2

3. Secondary Outcome: Adjusted Annualized Relapse Rate
Description: Clinical relapses are defined as new or recurrent neurologic symptoms, not associated with fever or infection, lasting for at least 24 hours, and accompanied by new objective neurological findings upon examination by the neurologist. The annualized relapse rate is calculated overall as the total number of relapses experienced in the study divided by the number of days followed in the study, and the ratio multiplied by 365. Obtained from a Poisson regression model, adjusted for the baseline relapse rate from study 101MS203 (NCT01440101).
Time Frame: Day 1 up to approximately 50 months
Measure: Number (95% Confidence Interval); unit: relapses per subject-years
Units Other Than Participants: Participants with a relapse
Arm/Group | Natalizumab
Number analyzed (Participants) | 97
Number analyzed (Participants with a relapse) | 26
relapses per subject-years | 0.243 [0.145 to 0.406]

4. Secondary Outcome: Mean Change From Baseline in the Assessment of Expanded Disability Status Scale (EDSS) up to Week 192
Description: The EDSS measures disability status on a scale ranging from 0 to 10, with higher scores indicating more disability. Scoring is based on measures of impairment in eight functional systems on examination by a neurologist.
Time Frame: Day 1 up to Week 192
Population: n=number of participants with an assessment at given timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Natalizumab
Number analyzed (Participants) | 97
units on a scale
  Change from Baseline to Week 12; n=92 | -0.05 (0.486)
  Change from Baseline to Week 24; n=86 | -0.15 (0.490)
  Change from Baseline to Week 36; n=84 | -0.08 (0.647)
  Change from Baseline to Week 48; n=78 | -0.09 (0.585)
  Change from Baseline to Week 60; n=76 | -0.09 (0.534)
  Change from Baseline to Week 72; n=72 | -0.04 (0.804)
  Change from Baseline to Week 84; n=60 | -0.08 (0.764)
  Change from Baseline to Week 96; n=53 | -0.10 (0.743)
  Change from Baseline to Week 108; n=46 | -0.18 (0.791)
  Change from Baseline to Week 120; n=38 | -0.12 (0.842)
  Change from Baseline to Week 132; n=31 | -0.11 (0.854)
  Change from Baseline to Week 144; n=22 | -0.07 (0.877)
  Change from Baseline to Week 156; n=11 | 0.14 (0.778)
  Change from Baseline to Week 168; n=8 | 0.31 (0.961)
  Change from Baseline to Week 180; n=8 | 0.25 (0.926)
  Change from Baseline to Week 192; n=2 | 0.50 (0.00)
  Change from Baseline to Final Treatment Visit;n=36 | -0.17 (0.862)

ADVERSE EVENTS:
Time Frame: Day 1 through First Follow-Up (12 Weeks After Last Infusion) +/- 7 days. Approximately 62 months.
Arm/Group | Natalizumab
Serious Adverse Events (participants affected / at risk) | 29/97
Other Adverse Events (participants affected / at risk) | 78/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Natalizumab (N=97)
Eosinophilia (Blood and lymphatic system disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Enteritis (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Oesophageal ulcer (Gastrointestinal disorders) | 1
Bronchitis (Infections and infestations) | 1
Meningitis (Infections and infestations) | 2
Mycoplasma infection (Infections and infestations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Central nervous system lesion (Nervous system disorders) | 1
Multiple sclerosis relapse (Nervous system disorders) | 17
Trigeminal neuralgia (Nervous system disorders) | 1
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
Asperger's disorder (Psychiatric disorders) | 1
Schizophrenia (Psychiatric disorders) | 1
Uterine prolapse (Reproductive system and breast disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Natalizumab (N=97)
Constipation (Gastrointestinal disorders) | 7
Dental caries (Gastrointestinal disorders) | 6
Diarrhoea (Gastrointestinal disorders) | 8
Gastritis (Gastrointestinal disorders) | 5
Stomatitis (Gastrointestinal disorders) | 5
Pyrexia (General disorders) | 6
Seasonal allergy (Immune system disorders) | 6
Cystitis (Infections and infestations) | 5
Gastroenteritis (Infections and infestations) | 5
Influenza (Infections and infestations) | 12
Nasopharyngitis (Infections and infestations) | 49
Pharyngitis (Infections and infestations) | 8
Fall (Injury, poisoning and procedural complications) | 5
Dizziness (Nervous system disorders) | 5
Headache (Nervous system disorders) | 6
Multiple sclerosis relapse (Nervous system disorders) | 21
Depression (Psychiatric disorders) | 5
Insomnia (Psychiatric disorders) | 10
Eczema (Skin and subcutaneous tissue disorders) | 8
Rash (Skin and subcutaneous tissue disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.